CLINICAL TRIAL: NCT02245503
Title: Comorbidity and Comedication During Prescription of ALNA® (Tamsulosin) for Patients With BPH (Benign Prostatic Hyperplasia)
Brief Title: Observational Study of ALNA® (Tamsulosin) in Patients With Benign Prostatic Hyperplasia (BPH)
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 527.40
Record Dates: First submitted 2014-09-18; First posted 2014-09-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Tamsulosin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Benign prostatic hyperplasia: Patients with symptomatic BPH to whom ALNA was prescribed
  Interventions: Drug: Tamsulosin

INTERVENTIONS:
Drug: Tamsulosin
  Other Names: ALNA

SUMMARY:
The objectives of this post marketing surveillance study were to document the comorbidity and comedication during prescription of ALNA® (Tamsulosin) for patients with BPH (Benign Prostatic Hyperplasia).

ELIGIBILITY:
Inclusion Criteria:

* Indication for the treatment with ALNA according to its summary of product characteristics (SPC)

Exclusion Criteria:

* Patients fulfilling one of the general or specific contraindications listed in the ALNA SPC, particularly patients with known hypersensitivities against tamsulosin hydrochloride or any other ingredient of the product, orthostatic dysregulation or severe liver insufficiency cannot be included in the study

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with BPH recruited at urologist offices
Sampling Method: Non-Probability Sample
Enrollment: 7391 (Actual)
Dates: Start 2003-05; Primary Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Collection of information on concomitant diseases | day 1
Collection of information on concomitant treatment | day 1

SECONDARY OUTCOMES:
Number of patients with adverse drug reactions | up to 6 months